CLINICAL TRIAL: NCT05750849
Title: Impact of Serum Progesterone Levels on the Day of β-hCG Test in Artificial Cycles on the Ongoing Pregnancy Rate.
Acronym: P4-BETA
Status: Recruiting | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 2209-VLC-135-EL
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Infertility, Female
Keywords: SERUM PROGESTERONE; LATE LUETEAL PHASE; ONGOING PREGNANCY RATE; ARTIFICIAL CYCLE; LUTEAL PHASE SUPPORT; EMBRYO TRANSFER
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OPTIMAL SERUM P4 LEVEL: Serum progesterone levels on β-hCG day over the threshold point calculated
  Interventions: Procedure: BLOOD COLLECTION FOR P4 DETERMINATION
- SUB-OPTIMAL SERUM P4 LEVEL: Serum progesterone levels on β-hCG day below the threshold point calculated
  Interventions: Procedure: BLOOD COLLECTION FOR P4 DETERMINATION

INTERVENTIONS:
Procedure: BLOOD COLLECTION FOR P4 DETERMINATION — Serum progesterone levels on the pregnancy test day

SUMMARY:
Prospective cohort multicentric study including infertile patients undergoing a pregnancy test on βhCG day (around ET +11), after an ET in the context of an artificial cycle and receiving LPS with vaginal natural progesterone following the clinical practice in IVI RMA (Spain).

DETAILED DESCRIPTION:
The investigation team have already demonstrated that serum progesterone levels measured on the ET day in artificial cycles are related to pregnancy outcome. In this line, this problem can be countteracted after supplementation with an additional source of external progesterone, achieving similar ongoing pregnancy and live birth rates in women with serum progesterone levels below and above the threshold point determined on the ET day.

Despite this, it has been observed apparent differences on the maintenance of pregnancy in patients with a positive pregnancy test according to their serum progesterone levels measured on day ET+11, which is the same day in which we perform the pregnancy test. These differences seem to be originated due to later higher clinical miscarriage rates in patients with lower serum progesterone levels on day ET+11, despite their positive pregnancy test.

This fact may be due to patientes low serum progesterone levels, insufficient to maintain an ongoing pregnancy. Taking this into account, this study aim to confirm that serum progesterone levels on βhCG day are indeed related to final pregnancy outcome and to evaluate if there is any cut-off point of serum progesterone levels, as we have previously found on the ET day.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent prior to any study related procedures
* Women ≤50 years old
* BMI ≤ 35 kg/m2
* Adequate endometrial thickness (>6.5mm) and pattern (Triple A structure) in the proliferative phase

Exclusion Criteria:

* Uterine Pathology, adnexal pathology
* Systemic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All infertile patients undergoing an embryo transfer in the context of an artificial cycle will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
LIVE BIRTH | 1 YEAR
  Record of live birth existence
ONGOING PREGNANCY | 1 YEAR
  Pregnancy confirmation by the observation of the presence of at least one gestational sac on ultrasound
POSITIVE PREGANCY | 1 YEAR
  Measurement of pregnancy test results
BIOCHEMICAL MISCARRIAGE | 1 YEAR
  Measurement of existence of miscarriage after a positive pregnancy test
CLINICAL MISCARRIAGE | 1 YEAR
  Measurement of existence of Miscarriage after confirmation of at least one gestational sac on ultrasound

SECONDARY OUTCOMES:
SERUM P4 LEVEL ON B-HCG DAY | 1 YEAR
  Measurement of serum progesterone levels on the pregnancy test day

CONTACTS AND LOCATIONS:
Locations (1):
- IVI RMA Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Labarta E, Rodriguez-Varela C, Mariani G, Bosch E. Serum Progesterone Profile Across the Mid and Late Luteal Phase in Artificial Cycles Is Associated With Pregnancy Outcome. Front Endocrinol (Lausanne). 2021 Jun 10;12:665717. doi: 10.3389/fendo.2021.665717. eCollection 2021. PMID 34177806